CLINICAL TRIAL: NCT01768416
Title: Measuring Depth of Unconsciousness at the End of Life: the Reliability of the BIS Monitoring as an Assessment Tool Versus Sedation Scales
Brief Title: Measuring Depth of Unconsciousness at the End of Life Using Bispectral Index (BIS)
Acronym: BISSOPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/895
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Loss of Consciousness at End of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to use the BIS monitor to assess the degree of consciousness in pre-terminal palliative patients admitted to our palliative care unit and to ascertain if this tool provides a more accurate assessment of consciousness in this specific group of patients than clinical observation of consciousness and the use of sedation scales.

We hypothesize that the measured BIS results provide a more accurate assessment of the patient's level of consciousness than routine clinical observation or the use of sedation scales.

ELIGIBILITY:
Inclusion Criteria:

* Pre-terminal palliative patients with a life expectancy of 72 hours or less at the start of the observation.

Exclusion Criteria:

* lack of consent of patient or representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-terminal palliative patients
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2015-09-23 (Actual); Study Completion 2015-09-23 (Actual)

PRIMARY OUTCOMES:
Measuring the accuracy of BIS monitoring in assessing the evolution of the level of consciousness in pre-terminal patients | 72 hours
  Measuring the accuracy of BIS monitoring in assessing the evolution of the level of consciousness in pre-terminal patients with a life expectancy of 72 hours or less from the moment of the first clinical signs of dying and loss of consciousness until the moment of death.

SECONDARY OUTCOMES:
Determining the evolution of BIS values, measured in pre-terminal patients | 72 hours
  Determining the evolution of BIS values, measured in pre-terminal patients with a life expectancy of 72 hours or less from the moment of the first clinical signs of dying and loss of consciousness until the moment of death.

OTHER OUTCOMES:
Determining the evolution of sedation scores, measured with the Observer's Assessment of Alertness/Sedation scale and the Richmond Agitation and Sedation Scale in pre-terminal patients | 72 hours
  Determining the evolution of sedation scores, measured with the Observer's Assessment of Alertness/Sedation scale and the Richmond Agitation and Sedation Scale in pre-terminal patients admitted to a palliative care unit with a life expectancy of 72 hours or less.
Determining if and in what degree the measured BIS values correspond to the measured sedation scores. | 72 hours
Determining if there is a noticeable difference between the BIS scores and sedation scale scores of patients with medically induced sedation | 72 hours
  Determining if there is a noticeable difference between the BIS scores and sedation scale scores of patients with medically induced sedation and those of patients losing consciousness as part of a normal dying process.

CONTACTS AND LOCATIONS:
Overall Officials: Martine De Laat, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium